CLINICAL TRIAL: NCT05605886
Title: The Effect of Botulinum Toxin A in Patients With Myofascial Pain Dysfunction Syndrome With and Without Zinc Supplementation (Randomized Controlled Trial)
Brief Title: Botulinum Toxin A in Patients With Myofascial Pain Syndrome With and Without Zinc Supplementation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Salah Fouad, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: botox in myofacial pain
Record Dates: First submitted 2022-09-29; First posted 2022-11-04 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Myofacial Pain Syndrome; Botulinum Toxin
MeSH Terms: conditions — Facial Neuralgia

STUDY DESIGN:
Intervention Model Description: All patients involved in this study will be divided in to two different groups, one group will undergo zinc supplement then botulinum toxins injection in masseter and temporalis muscle while the other group will have botulinum toxins injection in masseter and temporalis muscle without previous zinc supplement
Who Masked: Participant, Outcomes Assessor
Masking Description: 2 Cards will have sequential numbers one number for each card then these cards will be placed within opaque sealed envelopes. Then these envelops will be placed in a container (box), each participant will grasp one envelop the day of procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first group: (Control group) (Placebo Comparator): 1. EMG will be performed for masseter & temporalis muscles at the diagnosis appointment.
  2. Patients will recieve a daily placebo tablet in the morning after breakfast for 4 days prior to injections.
  3. Patients will receive a one-time treatment of 50 units of BoNT-A, the dose will be injected into the bilateral masseter muscles (16.7 units each masseter) and 1/3 into the bilateral temporalis (8.3 units each temporalis).
  4. Follow up will be performed using EMG for the masseter and temporalis muscles 4 months after the BoNT-A injection.
  Interventions: Drug: placebo
- second group. (intervention group) (Active Comparator): 1. EMG will be performed for masseter & temporalis muscles at the diagnosis appointment.
  2. Patients will receive a daily zinc supplement tablets of 50 mg in the morning after breakfast for 4 days prior to injections.
  3. Patients will receive a one-time treatment of 50 units of BoNT-A, the dose will be injected into the bilateral masseter muscles (16.7 units each masseter) and 1/3 into the bilateral temporalis (8.3 units each temporalis).
  4. Follow up will be performed using EMG for the masseter and temporalis muscles 4 months after the BoNT-A injection.
  Interventions: Drug: Solvazinc 50mg

INTERVENTIONS:
Drug: Solvazinc 50mg — Patients will receive a daily zinc supplement tablets of 50 mg in the morning after breakfast for 4 days prior to injections.
  Other Names: zinc supplement
  Arms: second group. (intervention group)
Drug: placebo — placebo
  Arms: first group: (Control group)

SUMMARY:
Research question:

Dose the use of oral zinc supplement improve the effects of botulinum toxins injection in patients with myofascial pain dysfunction syndrome?

Statement of the problem:

MPDS Patients treated with botulinum toxin A injection usually suffers from return of the symptoms which requires successive injections almost every (3-4M)

Rationale for conducting the research:

The concept of adding the zinc supplementation prior to BTXA injection is contributed to the fact that botulinum toxin is a zinc-dependent metalloprotease; therefore, every botulinum toxin molecule must be accompanied with a zinc molecule to effectively paralyze a muscle. However, commercially available BTXA preparations exclude zinc from their preparations, and BTX clinical efficiency and duration varies according to the zinc levels of the patient.

Although the BTX effect could remain for several months, its zinc-dependent proteolytic activity befalls within hours of administration before the toxins are degraded in the tissues.

Therefore, for achieving better results from BTX, the recipients should have adequate zinc levels at the time of administration. Therefore, oral zinc supplement intake prior to BTXA injection may enhance its clinical efficiency and duration.

botulinum neurotoxins are the most potent toxins known. They bind to nerve cells, penetrate the cytosol and block neurotransmitter release. Comparison of their predicted amino acid sequences reveals a highly conserved segment that contains the HExxH zinc binding motif of metalloendo peptidases. The metal content of tetanus toxin was then measured and it was found that one atom of zinc is bound to the light chain of tetanus toxin. Zinc could be reversibly removed by incubation with heavy metal chelators. Zn2+ is coordinated by two histidines with no involvement in cysteines, suggesting that it plays a catalytic rather than a structural role.

Bound Zn + was found to be essential for the tetanus toxin inhibition of neurotransmitter release in Aplysia neurons injected with the light chain. The intracellular activity of the toxin was blocked by phosphoramidon, a very specific inhibitor of zinc endopeptidases. Purified preparations of light chain showed a highly specific proteolytic activity against synaptobrevin, an integral membrane protein of small synaptic vesicles. The present findings indicate that tetanus toxin, and possibly also the botulinum neurotoxins, are metalloproteases and that they block neurotransmitter release via this protease activity. So The use of zinc supplementation prior to BTXA injection has been suggested by several previous studies to prolong its duration of action as well as improve its efficacy

DETAILED DESCRIPTION:
Myofascial pain syndrome is a complex disorder of the musculoskeletal system with multifactorial involvement and diverse clinical presentations in several areas of the body It can affect the oro-cranio-facial region, with involvement of the temporomandibular area and masticatory muscles, and is then called myofascial pain dysfunction syndrome.

Botulinum injections can improve blood flow to the muscles and release the nerve fibers compressed by abnormally contracting muscles, both of which may contribute to the cause of pain. In addition, botulinum injections can have an immediate effect owing to direct release of endogenous endorphins from introduction of the needle and alteration in the balance of central neurotransmitters; this is caused by local inhibition of pain peptides from sensory ganglions and nerve terminals, and anti-inflammatory and antiglutaminergic actions . Moreover, studies have shown that 3-10% of patients develop neutralizing antibodies with long-term adverse effects that include muscular atrophy.

BTX clinical efficiency and duration varies according to the zinc levels of the patient.

Although the BTX effect could remain for several months, its zinc-dependent proteolytic activity befalls within hours of administration before the toxins are degraded in the tissues.

Therefore, for achieving better results from BTX, the recipients should have adequate zinc levels at the time of administration. Therefore, oral zinc supplement intake prior to BTXA injection may enhance its clinical efficiency and duration.

Explanation for choice of comparators:

BTX is offered as a solution for myofascial pain patients; nevertheless, it is not considered as a definitive long-term solution so we add the zinc supplementation prior to BTXA injection to increase the clinical duration as reviewed in literature review.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myofascial pain
* Both genders males and females will be included.
* Ages from 17:50 Y
* General good health
* With complete dentation

Exclusion Criteria:

* Subjected to irradiation in the head and neck area less than 1 year ago
* Edentulous patients
* Patient with recent trauma.
* Poor motivation.
* Active infection area related to masseter or temporalis.
* Patient with anti-tetanus vaccine 1-3 m before experiment

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Muscular Activity | 4 months
  will be assessed by EMG
Pressure Pain Threshold (PPT) | 4 months
  will be assessed by algometer

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Galal, Study Director — professor; Omnia Adel aziz, Study Director — professor
Locations (1):
- Faculty of Dentistry, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen JL. Scientific skepticism and new discoveries: an analysis of a report of zinc/phytase supplementation and the efficacy of botulinum toxins in treating cosmetic facial rhytides, hemifacial spasm and benign essential blepharospasm. J Cosmet Laser Ther. 2014 Oct;16(5):258-62. doi: 10.3109/14764172.2014.948882. Epub 2014 Sep 2. PMID 25105993
- [Background] Lebeda FJ, Cer RZ, Mudunuri U, Stephens R, Singh BR, Adler M. The zinc-dependent protease activity of the botulinum neurotoxins. Toxins (Basel). 2010 May;2(5):978-97. doi: 10.3390/toxins2050978. Epub 2010 May 7. PMID 22069621
- [Background] Schiavo G, Poulain B, Rossetto O, Benfenati F, Tauc L, Montecucco C. Tetanus toxin is a zinc protein and its inhibition of neurotransmitter release and protease activity depend on zinc. EMBO J. 1992 Oct;11(10):3577-83. doi: 10.1002/j.1460-2075.1992.tb05441.x. PMID 1396558
- [Background] DE LA Torre Canales G, Camara-Souza MB, Poluha RL, Grillo CM, Conti PCR, Sousa MDLR, Rodrigues Garcia RCM, Rizzatti-Barbosa CM. Botulinum toxin type A and acupuncture for masticatory myofascial pain: a randomized clinical trial. J Appl Oral Sci. 2021 Jun 4;29:e20201035. doi: 10.1590/1678-7757-2020-1035. eCollection 2021. PMID 34105695